CLINICAL TRIAL: NCT03386617
Title: Open Label Single Arm Study for NEPA [oral Fixed-dose Combination of 300 Mg Netupitant and 0.50 Mg Palonosetron] in Hong Kong Oncology Patients Receiving (neo)-adjuvant Chemotherapy Treatment Consists of Adriamycin and Cyclophosphamide for Breast Cancer
Brief Title: AKY15-HK-301_NEPA Study
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Princess Margaret Hospital, Hong Kong (Other Government)
Responsible Party: Principal Investigator, CCTU, Principal Investigator, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYM011
Record Dates: First submitted 2017-11-22; First posted 2017-12-29 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NEPA (Experimental): Day 1 of each chemotherapy cycle:
  1 tablet of NEPA (NETU 300 mg/ PALO 0.50 mg) 1 hour prior to the start of chemotherapy with dexamethasone 12 mg administered orally 30 minutes prior to chemotherapy Days 2 to 3 Dexamethasone. The time and date of intake will be recorded.
  Interventions: Drug: NEPA

INTERVENTIONS:
Drug: NEPA — Day 1 of each chemotherapy cycle:
  1 tablet of NEPA (NETU 300 mg/ PALO 0.50 mg) 1 hour prior to the start of chemotherapy with dexamethasone 12 mg administered orally 30 minutes prior to chemotherapy Days 2 to 3 Dexamethasone. The time and date of intake will be recorded.

SUMMARY:
Nausea and vomiting (feeling sick to your stomach and throwing up) are two of the most common unpleasant side effects of chemotherapy agents (drugs specifically used to treat cancer) that will be used for cancer treatment. If nausea and vomiting are not controlled, they could lead to dehydration, poor nutrition and a longer time in the hospital. Nausea and vomiting usually occur in response to conditions that affect the gut and the vomiting center, which is an area in the brain.

Netupitant and palonosetron are drugs that are thought to block the activation of certain types of chemicals in these areas (brain and gut) and, therefore, to prevent or reduce the severity of nausea and vomiting. Nausea and vomiting caused by chemotherapy is classified into two patterns based on the time of onset or start. Acute nausea and vomiting start within 24 hours of chemotherapy administration. Delayed nausea and vomiting starts approximately 2-5 days after chemotherapy administration. Regardless of when the nausea and vomiting start, these symptoms are usually treated with not just one drug, but a combination of drugs. In this study you will receive the study drug, which is a fixed combination of netupitant and palonosetron.

This is an open label single arm study. The main purpose of this study or clinical trial is to learn more about the effect (how well it works) of the fixed combination of netupitant and palonosetron (NEPA) in preventing nausea and vomiting associated with chemotherapy in Hong Kong oncology patients receiving (neo)-adjuvant chemotherapy treatment consists of adriamycin and cyclophosphamide for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ( ≥ 18 and <75 years), female; a. Chinese patient, female ≥18 and < 75 years of age.
* Patient is diagnosed with early breast cancer.
* Patient is scheduled to receive her first course of (neo)- adjuvant chemotherapy for breast cancer follows:
* IV adriamycin 60 mg/m2 + cyclophosphamide 600 mg/m2
* ECOG Performance Status of 0-1;
* Written informed consent before study entry;
* If women of childbearing potential age: reliable contraceptive measures are to be used during all the planned course of the study;
* Ability and willingness of the patient to complete the diary and study questionnaires.

Exclusion Criteria:

* Any investigational drugs taken within 4 weeks prior to Day 1 of cycle 1, and/or is scheduled to receive any investigational drug during the study;
* Patients who are scheduled to receive concurrent radiation as part of their chemotherapy regimen for their malignancy;
* Patients who experience any vomiting or grade 2-3 nausea per Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v 4.03) in the 24 hours before Day 1 of chemotherapy;
* Patients who have taken any of the following agents within 7 calendar days prior to initiation of their chemotherapy regimen: 5-HT3 receptor antagonists, phenothiazines, benzamides, cannabinoids, NK1 receptor antagonists, corticosteroids, or benzodiazepines;
* Pregnant or breast-feeding women;
* Patient's inability to take oral medication;
* Gastrointestinal obstruction or active peptic ulcer;
* Psychiatric or CNS disorders interfering with ability to comply with study protocol;
* Patients at risk for severe cardiac/cardiovascular disorders
* Patients with myocardial infarction within 6 months

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the proportion of patients with a Complete Response (CR), during the delayed phase (24-120 h post-chemotherapy) periods in cycle 1 by using patient diary | up to 84 days
To evaluate the proportion of patients with Complete Protection during the delayed phase (24-120 h post-chemotherapy) periods in cycle 1 by using patient diary | up to 84 days

SECONDARY OUTCOMES:
Complete Response during the acute (0-24 h) phase in Cycle 1 by using patient diary | 6 days for every 3 weekly cycles. total 4 cycles, so time frame is 84 days
Complete Response during the overall (0-120 h) phase in Cycle 1 by using patient diary | 6 days for every 3 weekly cycles. total 4 cycles, so time frame is 84 days
Complete Protection during the acute (0-24 h) phase in Cycle 1 by using patient diary | 6 days for every 3 weekly cycles. total 4 cycles, so time frame is 84 days
Complete Protection during the overall (0-120 h) phase in Cycle 1 by using patient diary | 6 days for every 3 weekly cycles. total 4 cycles, so time frame is 84 days
Total Control during the acute, delayed and overall phases of Cycle 1; The percentage of patients with Total Control during the acute delayed phase in cycle 1 will be summarized descriptively | 6 days for every 3 weekly cycles. total 4 cycles, so time frame is 84 days
Total Control during the acute, delayed and overall phases of Cycle 1; The percentage of patients with Total Control during overall phase in cycle 1 will be summarized descriptively | 6 days for every 3 weekly cycles. total 4 cycles, so time frame is 84 days
Healthcare resources utilization; The number of hospitalizations will be summarized descriptively | 6 days for every 3 weekly cycles. total 4 cycles, so time frame is 84 days
Evaluation of NEPA safety profile; Clinical evaluations for safety assessments will include monitoring AEs | 6 days for every 3 weekly cycles. total 4 cycles, so time frame is 84 days
To assess the impact of nausea and vomiting on patients' quality of life, the FILE (Functional Living Index-Emesis) with a 5-day recall will be used. | 6 days for every 3 weekly cycles. total 4 cycles, so time frame is 84 days
A total FLIE score (expressed in FLIE points) greater than 108 will be categorized as having no impact on daily life | 6 days for every 3 weekly cycles. total 4 cycles, so time frame is 84 days

CONTACTS AND LOCATIONS:
Overall Officials: Winnie Yeo, MD, FRCP, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Clinical Oncology, Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yeo W, Lau TK, Kwok CC, Lai KT, Chan VT, Li L, Chan V, Wong A, Soo WM, Yeung EW, Wong KH, Tang NL, Suen JJ, Mo FK. NEPA efficacy and tolerability during (neo)adjuvant breast cancer chemotherapy with cyclophosphamide and doxorubicin. BMJ Support Palliat Care. 2022 Jul;12(e2):e264-e270. doi: 10.1136/bmjspcare-2019-002037. Epub 2020 Jan 29. PMID 31996363